CLINICAL TRIAL: NCT07372859
Title: Women's Heart: Impact of Ultra-endurance and Hormonal Profile on Cardiac and Systemic Inflammatory Parameters in Female Runners
Acronym: COEUR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-01
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: ultra endurance
MeSH Terms: interventions — Blood Specimen Collection; Weights and Measures; Surveys and Questionnaires; Antibody-Coated Bacteria Test, Urinary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will undergo examination before the race, during the race, at the arrival of the race, and 9 days after the race.
  Interventions: Procedure: Echocardiography; Procedure: Arterial ultrasound; Biological: Blood sampling; Behavioral: Scales and questionnaire; Procedure: Vital signs; Biological: Urinary test

INTERVENTIONS:
Procedure: Echocardiography — 6 transthoracic echocardiography will be performed: 1 before the race, 3 during the race (refreshment station), 1 at the end of the race, 1 at the follow up visit 9 days after the race. It is not possible to specify the intervention time, as this depends on the participants' running pace.
Procedure: Arterial ultrasound — 6 ultrasound of the carotid and femoral arteries will be performed: 1 before the race, 3 during the race (refreshment station), 1 at the end of the race, 1 at the follow up visit 9 days after the race. It is not possible to specify the intervention time, as this depends on the participants' running pace.
Biological: Blood sampling — 6 blood sampling (2 milliliters) will be performed: 1 before the race, 3 during the race (refreshment station), 1 at the end of the race, 1 at the follow up visit 9 days after the race. It is not possible to specify the intervention time, as this depends on the participants' running pace.
Behavioral: Scales and questionnaire — Before the race, during the race (refreshment station), and at the end of the race participant will be asked to complete the study questionnaire and scales. It is not possible to specify the intervention time, as this depends on the participants' running pace.
Procedure: Vital signs — 6 measurements of blood pressure, heart rate, respiratory rate, pulse oxygen saturation, and muscle oxygen saturation will then be taken: 1 before the race, 3 during the race (refreshment station), 1 at the end of the race, 1 at the follow up visit 9 days after the race. It is not possible to specify the intervention time, as this depends on the participants' running pace.
Biological: Urinary test — Pregnancy test will be performed before the race.

SUMMARY:
The goal of this clinical trial is to describe the cardiac and systemic inflammatory adaptations specific to women practicing ultra-endurance sports.

The objectives are to:

* Improve the understanding of cardiac and systemic inflammatory adaptations specific to women participating in ultra-endurance sports.
* Assess the relationship between observed cardiac and systemic inflammatory alterations and the relative levels of estrogen, testosterone, and progesterone.
* Describe the vascular adaptations specific to women participating in ultra-endurance sports.
* Examine the influence of defense mechanisms on the emotional dynamics observed during and after an ultra-endurance race.

DETAILED DESCRIPTION:
This is a French national non-comparative descriptive study. The study is conducted on healthy volunteers. 80 to 100 patients will be included, half of the inclusions on the "Ecotrail de Paris Ile France©"( = a trail running race in the Paris region. It is not possible to translate; it is a registered trademark) the second half of the inclusions on the "6000D©" in Savoie.

ELIGIBILITY:
Inclusion Criteria:

* Must have a Global Positioning System watch during the race;
* Must participate in one of the following races:

  * "Ecotrail de Paris Ile France©" (=a trail running race in the Paris region, it is not possible to translate; it is a registered trademark) 80 kilometers;
  * Or "la 6000D©" 69 kilometers;
* Must comply with the race regulations:

  * Medical certificate stating no contraindications to competitive running, dated less than 12 months prior to the race;
  * Or a valid sports license on the day of the race.
* Must agree to participate in the study, sign the consent form, and allow the sponsor to use their data for the purposes of this study.

Exclusion Criteria:

* Refusal or linguistic or mental incapacity to sign the informed consent form;
* Person under guardianship (conservatorship, curators, or legal protection) or deprived of liberty;
* Person not affiliated with a social security scheme;
* Pregnant woman;
* Person participating in a drug study;
* Women with a medical history (chronic lung disease, heart disease, pharmacologically treated hypertension) or with a known significant chronic inflammatory disease at the time of the enrollment visit;
* Person who has already participated in this study in a previous race.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-22 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac function | Before the race, at the 3 refreshment stations, at the arrival of the race, 9 days after the race.
  Echocardiographic measurements of left ventricular ejection fraction as a percentage
Systemic inflammatory parameters | Before the race, at the 3 refreshment stations, at the arrival of the race, 9 days after the race.
  Inflammatory profile adjusted for baseline

SECONDARY OUTCOMES:
Hormonal parameters | Before the race, at the 3 refreshment stations, at the arrival of the race, 9 days after the race.
  Hormonal profile adjusted for baseline
Vascular adaptations | Before the race, at the 3 refreshment stations, at the arrival of the race, 9 days after the race.
  Carotid artery and femoral artery diameter adjusted for baseline
Defense mechanisms regarding emotional dynamics | Before the race, at the 3 refreshment stations, at the arrival of the race.
  Defense Style Questionnaire-26 questionnaire is a standardized questionnaire developed to assess defense mechanisms: adaptive (humor, anticipation, self-assertion, altruism, self-observation) and maladaptive defenses (help rejecting complaining, splitting other, projection, dissociation, intellectualization, devaluation/self, fantasy, devaluation of other). These items are rated on a Likert scale from 1 to 6 points; 1 corresponding to "strongly disagree" and 6 to "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Romain JOUFFROY, MD, Principal Investigator — CHU d'Orléans
Locations (1):
- Hôpital Henri Mondor, APHP, Créteil, France